CLINICAL TRIAL: NCT02491983
Title: A Randomized, Multicenter, Open-label, Phase II Trial to Evaluate the Efficacy and Safety of Palbociclib in Combination With Fulvestrant or Letrozole in Patients With HER2 Negative, ER+ Metastatic Breast Cancer
Brief Title: Palbociclib in Combination With Fulvestrant or Letrozole in Patients With ER+, HER2- Advanced Breast Cancer
Acronym: PARSIFAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP067; 2014-004698-17 (EudraCT Number)
Record Dates: First submitted 2015-06-29; First posted 2015-07-08 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; Endocrine receptors positive; HER-2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Combination of Palbociclib and Letrozole
  Interventions: Drug: Palbociclib; Drug: Letrozole
- Arm B (Experimental): Combination of Palbociclib and Fulvestrant
  Interventions: Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib
  Other Names: PD-0332991
Drug: Fulvestrant
  Other Names: Faslodex
  Arms: Arm B
Drug: Letrozole
  Other Names: Femara
  Arms: Arm A

SUMMARY:
This is an international, randomized, open-label, controlled, multicenter phase II clinical trial to investigate and compare the safety and efficacy of palbociclib combined with fulvestrant or letrozole in women with ER+, HER2- locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
Patients will be stratified by site of disease (visceral vs. non-visceral) and by onset of metastatic disease diagnose (patients metastatic de novo versus non de novo).

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older with metastatic or locally advanced disease, not amenable to curative therapy
2. Confirmed diagnosis of HR+/HER2- breast cancer
3. Post-menopausal status
4. No prior chemotherapy line in the metastatic setting
5. Measurable disease defined by RECIST version 1.1, or non-measurable disease
6. Eastern Cooperative Oncology Group (ECOG) PS 0-1
7. Adequate organ and marrow function, resolution of all toxic effects of prior therapy or surgical procedures
8. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCICTCAE version 4.0 Grade equal or minor than 1

Exclusion Criteria:

1. ER or HER2 unknown disease
2. HER2 positive disease based on local laboratory results
3. Locally advanced breast cancer candidate for a radical treatment
4. Prior (neo)adjuvant endocrine treatment with DFI ≤ 12-months from completion of treatment.
5. Patients with rapidly progressive visceral disease or visceral crisis.
6. Major surgery within 4 weeks of start of study drug
7. Patients with an active, bleeding diathesis
8. Serious concomitant systemic disorder incompatible with the study
9. Are unable to swallow tablets
10. Chronic daily treatment with corticosteroids with a dose of ≥ 10mg/day methylprednisolone equivalent
11. Known active uncontrolled or symptomatic CNS metastases
12. Known hypersensitivity to letrozole, fulvestrant or any of their excipients, or to any PD-0332991 excipients
13. QTc > 480 msec on basal assessments, personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes
14. Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, Principal Investigator — MedSIR
Locations (41):
- Czechia (2):
  - MedSIR investigative site, Olomouc
  - MedSIR investigative site, Prague
- France (3):
  - MedSIR investigative site, Paris
  - MedSIR investigative site, Strasbourg
  - MedSIR investigative site, Toulouse
- Germany (2):
  - MedSIR investigative site, Dessau
  - MedSIR investigative site, Heidelberg
- Italy (8):
  - MedSIR investigative site, Brindisi
  - MedSIR investigative site, Cagliari
  - MedSIR investigative site, Cremona
  - MedSIR investigative site, Milan
  - MedSIR investigative site, Modena
  - MedSIR investigative site, Monza
  - MedSIR investigative site, Piacenza
  - MedSIR investigative site, Torino
- Russia (3):
  - MedSIR investigative site, Moscow
  - MedSIR investigative site, Saint Petersburg
  - MedSIR investigative site, Yaroslavl
- Spain (16):
  - MedSIR investigative site, Barcelona
  - MedSIR investigative site, Bilbao
  - MedSIR investigative site, Castelló
  - MedSIR investigative site, Cáceres
  - MedSIR investigative site, Córdoba
  - MedSIR investigative site, Girona
  - MedSIR investigative site, Huelva
  - MedSIR investigative site, Madrid
  - MedSIR investigative site, Oviedo
  - MedSIR investigative site, Pamplona
  - MedSIR investigative site, Santiago de Compostela
  - MedSIR investigative site, Seville
  - MedSIR investigative site, Tarragona
  - MedSIR investigative site, Valencia
  - MedSIR investigative site B, Zaragoza
  - MedSIR investigative site, Zaragoza
- United Kingdom (7):
  - MedSIR investigative site, Bath
  - MedSIR investigative site, London
  - MedSIR investigative site, Manchester
  - MedSIR investigative site, Nottingham
  - MedSIR investigative site, Romford
  - MedSIR investigative site, Swansea
  - MedSIR investigative site, Truro

REFERENCES:
- [Derived] Di Cosimo S, Perez-Garcia JM, Bellet M, Dalenc F, Gil Gil MJ, Ruiz Borrego M, Gavila J, Sampayo-Cordero M, Aguirre E, Schmid P, Marme F, Gligorov J, Schneeweiss A, Albanell J, Zamora P, Wheatley D, Martinez-De Duenas E, Caranana V, Amillano K, Mina L, Malfettone A, Cortes J, Llombart-Cussac A. Palbociclib with Fulvestrant or Letrozole in Endocrine-Sensitive Patients with HR-Positive/HER2-Negative Advanced Breast Cancer: A Detailed Safety Analysis of the Randomized PARSIFAL Trial. Oncologist. 2023 Jan 18;28(1):23-32. doi: 10.1093/oncolo/oyac205. PMID 36239405
- [Derived] Llombart-Cussac A, Perez-Garcia JM, Bellet M, Dalenc F, Gil-Gil M, Ruiz-Borrego M, Gavila J, Sampayo-Cordero M, Aguirre E, Schmid P, Marme F, Di Cosimo S, Gligorov J, Schneeweiss A, Albanell J, Zamora P, Wheatley D, Martinez-de Duenas E, Amillano K, Malfettone A, Cortes J; PARSIFAL Steering Committee and Trial Investigators. Fulvestrant-Palbociclib vs Letrozole-Palbociclib as Initial Therapy for Endocrine-Sensitive, Hormone Receptor-Positive, ERBB2-Negative Advanced Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2021 Dec 1;7(12):1791-1799. doi: 10.1001/jamaoncol.2021.4301. PMID 34617955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women and premenopausal women receiving LHRH analogues, aged ≥ 18 years with ER+ and HER2- with laBC or mBC that had not received any therapy for the metastatic disease.
Pre-assignment Details: Screening details:
  * Postmenopausal and premenopausal women receiving LHRH analogues, ≥ 18 years.
  * ECOG score ≤ 2
  * Histologically confirmed ER+ and/or PgR+ and HER2- locally advanced or MBC
  * Not candidates for a local treatment with a radical intention
  * No prior therapy for metastatic disease.
  * Evidence of measurable or evaluable metastatic disease
Groups:
- Arm A: Combination of Palbociclib and Letrozole
  Palbociclib
  Letrozole
- Arm B: Combination of Palbociclib and Fulvestrant
  Palbociclib
  Fulvestrant
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 243 | 243
Completed | 241 | 242
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Not meet selection criteria | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 243 | 243 | 486
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 142 | 131 | 273
  >=65 years | 101 | 112 | 213
Age, Continuous [Median (Full Range); unit: years] | 62 [35 to 90] | 64 [25 to 88] | 63 [25 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243 | 243 | 486
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125 | 130 | 255
  Not Hispanic or Latino | 107 | 106 | 213
  Unknown or Not Reported | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 230 | 231 | 461
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  Czechia | 7 | 7 | 14
  Italy | 21 | 17 | 38
  United Kingdom | 29 | 25 | 54
  France | 34 | 36 | 70
  Germany | 11 | 13 | 24
  Russia | 16 | 15 | 31
  Spain | 125 | 130 | 255

OUTCOME MEASURES:

1. Primary Outcome: 1-year Progression Free Survival
Description: Percentage of patients who are alive and without evidence of tumor progression (defined using RECIST v1.1)
Time Frame: One year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 243 | 243
percentage of participants | 79.4 [73.6 to 84] | 77.9 [72 to 82.8]

2. Secondary Outcome: Number of Participants With Grade 3/4 Adverse Events, SAEs, Deaths and Discontinuations •
Description: Grade 3/4 adverse events, SAEs, deaths and discontinuations following the CTCAE v5 criteria
Time Frame: Through study completion. From baseline up to 51 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 243 | 243
Participants | 243 | 243

3. Secondary Outcome: Time To Progression (TTP)
Description: Time from randomization to disease progression
Time Frame: Through study completion. From baseline up to 51 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 243 | 243
months | 32.8 [26 to 38.6] | 28.9 [24.6 to 36.2]

4. Secondary Outcome: Overall Survival (OS)
Description: Time from date of randomization to date of death due to any cause
Time Frame: Through study completion. From baseline up to 51 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 243 | 243
months | NA [49.9 to NA] — There were not enough events to calculate the OS. 50% of the patients did not die. | NA [49 to NA] — There were not enough events to calculate the OS. 50% of the patients did not die.

5. Secondary Outcome: Clinical Benefit Rate
Description: Percentage of patients who experience a CR, PR or stable disease (for at least 24 weeks) and assessed by modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria.
Time Frame: Through study completion. From baseline up to 51 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 243 | 243
percentage of participants | 69.1 [62.9 to 74.9] | 70.8 [64.6 to 76.4]

6. Secondary Outcome: Overall Response Rate
Description: Proportion of patients with best overall response of confirmed complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST criteria guidelines (version 1.1)
Time Frame: Through study completion. From baseline up to 51 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 243 | 243
Participants | 112 | 106

ADVERSE EVENTS:
Time Frame: Through study completion. From baseline up to 51 months.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 2/243 | 8/243
Serious Adverse Events (participants affected / at risk) | 51/243 | 72/243
Other Adverse Events (participants affected / at risk) | 242/243 | 241/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=243) | Arm B (N=243)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Infections and infestations) | 2 (2) | 6 (6)
Severe asthma with fungal sensitisation (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Radiotherapy to bone (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal corpectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=243) | Arm B (N=243)
Neutropenia (Blood and lymphatic system disorders) | 207 (207) | 198 (198)
Lymphopenia (Blood and lymphatic system disorders) | 18 (18) | 18 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 39 (39) | 49 (49)
Leukopenia (Blood and lymphatic system disorders) | 61 (61) | 60 (60)
Anaemia (Blood and lymphatic system disorders) | 68 (68) | 55 (55)
Vertigo (Ear and labyrinth disorders) | 10 (10) | 13 (13)
Toothache (Gastrointestinal disorders) | 11 (11) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 12 (12) | 9 (9)
Haemorrhoids (Gastrointestinal disorders) | 13 (13) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 15 (15) | 18 (18)
Dyspepsia (Gastrointestinal disorders) | 25 (25) | 21 (21)
Abdominal pain upper (Gastrointestinal disorders) | 31 (31) | 22 (22)
Vomiting (Gastrointestinal disorders) | 39 (39) | 35 (35)
Constipation (Gastrointestinal disorders) | 40 (40) | 34 (34)
Nausea (Gastrointestinal disorders) | 45 (45) | 57 (57)
Stomatitis (Gastrointestinal disorders) | 48 (48) | 40 (40)
Diarrhoea (Gastrointestinal disorders) | 60 (60) | 65 (65)
Gastrointestinal disorders (Gastrointestinal disorders) | 158 (158) | 168 (168)
Injection site pain (General disorders) | 0 (0) | 15 (15)
Pain (General disorders) | 14 (14) | 16 (16)
Oedema peripheral (General disorders) | 22 (22) | 18 (18)
Pyrexia (General disorders) | 24 (24) | 23 (23)
Fatigue (General disorders) | 63 (63) | 62 (62)
Asthenia (General disorders) | 87 (87) | 90 (90)
Respiratory tract infection (Infections and infestations) | 7 (7) | 14 (14)
Conjunctivitis (Infections and infestations) | 11 (11) | 13 (13)
Pharyngitis (Infections and infestations) | 13 (13) | 4 (4)
Influenza (Infections and infestations) | 15 (15) | 20 (20)
Bronchitis (Infections and infestations) | 15 (15) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 15 (15)
Urinary tract infection (Infections and infestations) | 26 (26) | 23 (23)
Viral upper respiratory tract infection (Infections and infestations) | 32 (32) | 32 (32)
Aspartate aminotransferase increased (Investigations) | 15 (15) | 13 (13)
Alanine aminotransferase increased (Investigations) | 16 (16) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 33 (33) | 34 (34)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 12 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 15 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (16) | 11 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 19 (19) | 24 (24)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 (23) | 27 (27)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (28) | 39 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 49 (49) | 57 (57)
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 (80) | 62 (62)
Paraesthesia (Nervous system disorders) | 14 (14) | 17 (17)
Dysgeusia (Nervous system disorders) | 16 (16) | 13 (13)
Dizziness (Nervous system disorders) | 20 (20) | 16 (16)
Headache (Nervous system disorders) | 33 (33) | 34 (34)
Depression (Psychiatric disorders) | 10 (10) | 15 (15)
Anxiety (Psychiatric disorders) | 19 (19) | 11 (11)
Insomnia (Psychiatric disorders) | 21 (21) | 18 (18)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 12 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 14 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 33 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (42) | 54 (54)
Rash (Skin and subcutaneous tissue disorders) | 15 (15) | 26 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (19) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (25) | 28 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 61 (61) | 56 (56)
Hypertension (Vascular disorders) | 13 (13) | 10 (10)
Hot flush (Vascular disorders) | 46 (46) | 41 (41)

LIMITATIONS AND CAVEATS:
The number of deaths was not sufficient to determine the secondary objective of calculating Overall Survival, so this value could not be obtained. We consider the fact that we were not able to obtain this factor to be very positive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT02491983/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT02491983/SAP_001.pdf
  • Informed Consent Form (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT02491983/ICF_002.pdf